CLINICAL TRIAL: NCT01124006
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of 2 Doses of Intradiscal rhGDF-5 (Single Administration) for the Treatment of Early Stage Lumbar Disc Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-Intradiscal rhGDF-5-04
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Intradiscal rhGDF-5 (Experimental): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.
  Interventions: Drug: Intradiscal rhGDF-5
- Water for injection (Placebo Comparator): Sterile water for injection
  Interventions: Other: Water for injection

INTERVENTIONS:
Drug: Intradiscal rhGDF-5 — The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.
  Arms: Intradiscal rhGDF-5
Other: Water for injection — Sterile water for injection
  Arms: Water for injection

SUMMARY:
Study to show the safety and tolerability of Intradiscal rhGDF-5 in subjects with early lumbar disc degeneration

ELIGIBILITY:
Inclusion Criteria:

1. Persistent low back pain with at least 3 months of non-surgical therapy at one suspected symptomatic lumbar level (L3/L4 to L5/S1) as confirmed using a standardized provocative discography protocol. The required discography protocol will be provided by the sponsor. Subjects with multilevel disease must have a provocative discogram confirming that only 1 level is symptomatic at least 2 weeks prior to administration. Historical provocative discograms may be used for screening purposes, with an expiry of 12 calendar months from the date performed. If the study treatment is not performed within those 12 calendar months, a new discogram will be required.
2. Oswestry Disability Index (ODI) for low back pain of 30 or greater
3. Low Back Pain score greater than or equal to 4 cm as measured by Visual Analog Scale (VAS) at Visit 1 Baseline

Exclusion Criteria:

1. Persons unable to have a discogram, CT, or MRI
2. Abnormal neurological exam at baseline (e.g., chronic radiculopathy)
3. Active radicular pain due to anatomical compression such as stenosis or disc herniation (radicular pain is defined as pain below the knee)
4. Extravasation of contrast agent during the discogram, into the epidural space (does not include leakage of contrast agent along the needle track or leakage to the outer annular ring at the posterior longitudinal ligament vicinity)
5. Suspected symptomatic facet joints and/or severe facet joint degeneration at the index level or adjacent segments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Hope Research Institute, Phoenix, Arizona
  - The Spine Institute, Santa Monica, California
  - Durango Orthopedic Associates/Spine Colorado, Durango, Colorado
  - Drug Studies America, Marietta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hospital for Special Surgery, New York, New York
  - University Orthopedics Center, State College, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Spine Team Texas, Southlake, Texas
  - Texas Spine & Joint Hospital, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Intradiscal rhGDF-5 (1.0mg); Intradiscal rhGDF-5 (2.0mg): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc.
- Placebo: Excipients in Intradiscal rhGDF-5, to include Trehalose, Glycine, HCl, and Water for Injection
Period: Overall Study
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Started | 10 | 10 | 4
Completed | 7 | 8 | 2
Not Completed | 3 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg) | Total
Number analyzed (Participants) | 10 | 10 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (9.56) | 44.7 (7.86) | 42.4 (6.38) | 42.2 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 8
  Male | 6 | 7 | 3 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Neurological Assessment for Motor Function and Reflexes/Sensory
Description: Neurological Assessment for Motor Function and Reflexes/Sensory- Number of patients with Clinically Significant Abnormal results at 12 months.
  For Motor Function, Clinically Significant Abnormal results are determined by the surgeon investigator and are further classified by grade: 0= No Movement, 1= Flicker/trace of contraction, 2=Active movement when gravity removed, 3= Active movement against gravity, 4= Active Movement against gravity and resistance.
  For Reflexes/Sensory, Clinically Significant Abnormal results are determined by the surgeon investigator and are based on exams of the Knee, Ankle, L3-L5 Dermatone, and S1 Dermatome. Tension signs are evaluated with a straight leg raise to determine at which point, if any, sciatic pain occurs.
Time Frame: 12 months
Population: Safety Population
  For the Neurological Assessment at 12 months, only 8 subjects from the rhGDF-5 1.0mg group (out of 10 subjects total) completed the assessment, only 3 subjects from the rhGDF-5 2.0mg group (out of 4 subjects total) completed the assessment, and none of the placebo subjects (out of 10 total subjects) completed the assessment.
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 8 | 0 | 3
participants | 0 |  | 0

2. Secondary Outcome: Change in Function Assessed by Oswestry Disability Index Change at 12 Months From Baseline.
Description: The Oswestry Disability Index (ODI) is a 10-category (Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, Traveling) disability measurement scale with a graded response from 0 to 5, with 0 being the best score (no impairment) to 5 being the worst score (significant impairment). ODI score for a subject is calculated by adding the scores and converting the score to a 100 point scale.
Time Frame: 12-month
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 10 | 10 | 4
units on a scale | -19.8 (21.22) | -18.8 (22.43) | -6.0 (29.98)

3. Secondary Outcome: Change in Pain Visual Analogue Scale (VAS) at 12 Months From Baseline.
Description: The Visual Analogue Scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line ( that is approximately 10cm long) with 'No Pain' (score of 0=0cm) listed on the left and 'Very severe pain' (score of 10=10cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their back.
Time Frame: 12 months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 10 | 10 | 4
units on a scale | -2.33 (3.645) | -2.78 (3.751) | -1.10 (3.336)

4. Secondary Outcome: Change in Physical Component Summary of Quality of Life Measure Assessed by Short-Form 36 at 12 Months From Baseline.
Description: The 36-item Short Form Health Survey (SF-36) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into two summary measures (the Physical Component- PCS and Mental Component- MCS) that are scored from 0 to 100 (where 100 indicates the highest level of health)
Time Frame: 12 months
Population: FAS Population
  One subject from the rhGDF-5 1.0mg group (out of 10 subjects total) did not complete the PCS, SF-36 at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 9 | 10 | 4
units on a scale | 7.22 (9.728) | 8.61 (14.213) | 6.21 (8.245)

5. Secondary Outcome: Change in Mental Component Summary Quality of Life Measure Assessed by Short Form SF-36 at 12 Months From Baseline.
Description: as for outcome 4
Time Frame: 12 months
Population: FAS Population
  One subject from the rhGDF-5 1.0mg group (out of 10 subjects total) did not complete the MCS, SF-36 at Baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 9 | 10 | 4
units on a scale | 2.86 (11.142) | -0.92 (9.163) | 1.31 (20.276)

6. Primary Outcome: Treatment Emergent Adverse Events- Relationship to Study Drug
Description: Number of patients with Treatment Emergent Adverse Events that were designated as Definitely Related to Study Drug.
Time Frame: Through a 12 month period and annual telephone contact at 24 and 36 months for subject health status follow-up.
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 10 | 10 | 4
participants | 0 | 0 | 0

7. Primary Outcome: Treatment Emergent Adverse Events- Relationship to Study Drug
Description: Number of patients with Treatment Emergent Adverse Events that were designated as Possibly or Probably Related to Study Drug.
Time Frame: 12 month period and annual telephone contact at 24 and 36 months for subject health status follow-up
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 10 | 10 | 4
participants | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected through a 12 month period and annual telephone contact at 24 months and 36 months.
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Placebo | Intradiscal rhGDF-5 (2.0mg)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 2/4
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (1.0mg) (N=10) | Placebo (N=10) | Intradiscal rhGDF-5 (2.0mg) (N=4)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (1.0mg) (N=10) | Placebo (N=10) | Intradiscal rhGDF-5 (2.0mg) (N=4)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (18) | 6 (9) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 4 (5) | 0 (0) | 1 (1)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infections (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 3 (3) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Burning Sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood Cholesteral Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Urine Present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac Murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lasegue's Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Puritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Investigators may freely present or publish results of the Clinical Investigation in a manner which fairly sets forth the conclusions reached by the Clinical Investigators, but only after the Sponsor has been given the opportunity of reviewing the proposed presentation or publication at least 60 days prior to the intended submission, presentation, or publication date.